CLINICAL TRIAL: NCT04084340
Title: Efficacy of Transcranial Direct Current Stimulation Combined With Exercise Therapies in Female Urinary Incontinence: a Randomized Clinical Trial
Brief Title: tDCS and Female Urinary Incontinence
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Universidade Federal do Piauí (Other)
Responsible Party: Principal Investigator, Fuad Ahmad Hazime, Clinical Professor - Physical Therapy Department, Universidade Federal do Piauí
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: tDCS and Urinary Incontinence
Record Dates: First submitted 2019-09-02; First posted 2019-09-10 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence | interventions — Exercise Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anodal tDCS + Exercises therapies (Experimental): Real transcranial direct current stimulation associated with therapeutic exercises
  tDCS: 20 minutes, 2mA
  Interventions: Procedure: Real transcranial direct current stimulation + therapeutic exercises for urinary incontinence
- Sham tDCS + Exercises therapies (Sham Comparator): Sham transcranial direct current stimulation associated with therapeutic exercises
  tDCS: 20 minutes (30 seconds ON), 2mA
  Interventions: Procedure: Sham transcranial direct current stimulation + therapeutic exercises for urinary incontinence

INTERVENTIONS:
Procedure: Real transcranial direct current stimulation + therapeutic exercises for urinary incontinence — Real transcranial direct current stimulation associated with therapeutic exercises for urinary incontinence
  tDCS: 20 minutes, 2mA, motor supplementary area anode and supraorbital cathode (ipsilateral to the dominant lower limb).Technique based on the application of weak, direct electrical current to the brain through relatively large electrodes that are placed over the scalp, in which anodal and cathodal stimulation increases and decreases cortical excitability, respectively.
  Arms: Anodal tDCS + Exercises therapies
Procedure: Sham transcranial direct current stimulation + therapeutic exercises for urinary incontinence — Sham transcranial direct current stimulation + therapeutic exercises for urinary incontinence
  tDCS: 20 minutes (30 seconds ON), 2mA, motor supplementary area anode and supraorbital cathode (ipsilateral to the dominant lower limb).Technique based on the application of weak, direct electrical current to the brain through relatively large electrodes that are placed over the scalp, in which anodal and cathodal stimulation increases and decreases cortical excitability, respectively.
  Arms: Sham tDCS + Exercises therapies

SUMMARY:
Urinary incontinence (UI) is defined as any involuntary loss of urine and can be divided into three types: urgency, stress and mixed. Pelvic floor exercises are considered the main non pharmacological choice for UI treatment. Its mechanisms are not fully understood, however there are some evidence that central mechanisms play an important role in the continence control. In this context, neuromodulatory techniques, such as transcranial direct current stimulation (tDCS), that address cortical targets has been demonstrated promising results in different health conditions. However, few studies have investigated the efficacy of adding tDCS to exercise therapies for women with UI.

ELIGIBILITY:
Inclusion Criteria:

* Complaining of urinary loss
* Seeking care for urinary incontinence

Exclusion Criteria:

* Grade III vaginal dystopias
* Intrapelvic tumors
* Cardiac pacemaker or other implanted devices
* Current pregnancy
* Urinary tract infections
* Previous treatment with tDCS

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-11-14 (Actual); Primary Completion 2021-01-15 (Actual); Study Completion 2023-11-27 (Actual)

PRIMARY OUTCOMES:
Urinary leakage | 4 weeks after randomization
  Urinary leakage will be measured by the pad test. Pad testing yields an objective measurement of fluid loss over a certain period.
  The outcome of the 1-h pad test will be recorded as the weight gain as measured by a verified spring balance.
  Pad test assessment: Change in 1-hour exercise (stress), classified as mild, moderate or severe urinary leaking.
Incontinence severity | 4 weeks after randomization
  Incontinence severity will be assessed by the Brazilian version of Incontinence severity index (ISI) that quantifies the frequency and number of urinary leaking.
  The ISI comprehend two questions about quantity and frequency of urinary losses. The score are from 0 to 12:
  0 continent
  1 or 2 mild incontinence 3 or 6 moderate incontinence 8 or 9 severe incontinence 12 very severe incontinence
Quality of life impact | 4 weeks after randomization
  Quality of life impact of urinary incontinence will be assessed by the Brazilian Version of International consultation on incontinence questionnaire urinary incontinence (ICIQ_UI short form).
  The ICIQ-UI Short form provides a score ranging from 0-21. With a higher score indicating greater severity of symptoms.

SECONDARY OUTCOMES:
Urinary leakage | 3 and 6 months after randomization
  Urinary leakage will be measured by the pad test. Pad testing yields an objective measurement of fluid loss over a certain period.
  The outcome of the 1-h pad test will be recorded as the weight gain as measured by a verified spring balance.
  Pad test assessment: Change in 1-hour exercise (stress), classified as mild, moderate or severe urinary leaking.
Incontinence severity | 3 and 6 months after randomization ]
  Incontinence severity will be assessed by the Brazilian version of Incontinence severity index (ISI) that quantifies the frequency and number of urinary leaking.
  The ISI comprehend two questions about quantity and frequency of urinary losses. The score are from 0 to 12:
  0 continent
  1 or 2 mild incontinence 3 or 6 moderate incontinence 8 or 9 severe incontinence 12 very severe incontinence
Quality of life impact | 3 and 6 months after randomization ]
  Quality of life impact of urinary incontinence will be assessed by the Brazilian Version of International consultation on incontinence questionnaire urinary incontinence (ICIQ_UI short form).
  The ICIQ-UI Short form provides a score ranging from 0-21. With a higher score indicating greater severity of symptoms.
Quality of life in women with UI (severity symptoms) | 4 weeks, 3 and 6 months after randomization
  Quality of life will be analyzed by the Brazilian version of King's Health Questionnaire.
  KHQ is a patient self-administered self-report and has 3 parts consisting of 21 items. The score from eight subscales "domains" are from 0 (best) to 100 (worst). Decreases in KHQ domain scores indicate an improvement in quality of life.
Emotional impact | 4 weeks, 3 and 6 months after randomization
  The emotional impact of urinary incontinence on quality of life will be analyzed by the Brazilian version of Incontinence Quality of Life Questionnaire (IQOL) that evaluates the social, physical and mental aspects of the woman with urinary incontinence.
  The IQOL is a self-report questionnaire with 22 questions and three subscales ("domains"). The score are from 0 (worst) to 100 (best).
Pelvic floor muscle strength - Subjective test | 4 weeks, 3 and 6 months after randomization
  Pelvic floor strength will be analyzed by Bidigital vaginal palpation of the vaginal introitus.
Pelvic floor muscle strength - Quantitative test | 4 weeks, 3 and 6 months after randomization
  Pelvic floor strength will be analyzed by a clinical perineometer in cm H2O.
Urinary leaking | 4 weeks, 3 and 6 months after randomization
  Diary delivered to the participant to note for 24h the urinary frequency daytime, night, amount of loss and exchange of absorbents if you use.
Global perceived effect (GPE) | 4 weeks, 3 and 6 months after randomization
  Global perceived effect is an 11 point scale that ranges from 5 (vastly worse) through 0 (no change) to 5 (completely recovered).

OTHER OUTCOMES:
Depression | 4 weeks, 3 and 6 months after randomization
  Beck depression inventory (BDI) for depressive symptoms that we tracked as possible confounding factor.
  The BDI is a tool of self-assessment of depression using a questionnaire with 21 items whose in- tensity varies from 0 to 3 (higher scores indicating more depressive symptoms).
Anxiety | 4 weeks, 3 and 6 months after randomization
  Visual analogue scale (VAS) for anxiety assesses anxiety symptoms that we tracked as possible confounding factor.
  The visual analogue scale for general anxiety is assessed by a horizontal 100-mm-long line. The score are from 0 (worst) to 100 (best).
Satisfaction with care: Medrisk Instrument | 4 weeks after randomization
  Satisfaction with care will be measured by the Medrisk Instrument for Measuring Patient Satisfaction with Physiotherapy Care.

CONTACTS AND LOCATIONS:
Locations (2):
- Brazil (2):
  - Department of Physical Therapy. Federal University of Piaui, Parnaíba, Piauí
  - Antonia Mykaele Cordeiro Brandao, Parnaíba, Piauí

IPD SHARING:
Plan to Share IPD: No